CLINICAL TRIAL: NCT06116799
Title: Managing Pain in Patients With Plantar Fasciitis - A Blinded Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient power;slowed enrollment pace;budget restraints
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Soheil Ashkani Esfahani, Director, Foot and Ankle Research and Innovation Laboratory, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P003250
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Orthotic Devices

STUDY DESIGN:
Intervention Model Description: 19 patients with plantar fasciitis will be allocated to carbon fiber insole group 19 patients with plantar fasciitis will be allocated to polyurethane insole group 19 patients with plantar fasciitis will be allocated to polyethylene insole group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbon fiber insole (Experimental): assigned carbon fiber insole
  Interventions: Device: Orthotic
- Polyurethane (Active Comparator): Assigned polyurethane insole
  Interventions: Device: Orthotic
- Polyethylene (Active Comparator): assigned polyethylene insole
  Interventions: Device: Orthotic

INTERVENTIONS:
Device: Orthotic — Arch support orthotic

SUMMARY:
Plantar fasciitis (PF), a leading cause of persistent heel pain, results in almost a million physician visits annually. Conservative treatment is often the first line of management with insoles being frequently prescribed. While multiple studies have compared insoles based on the degree of customization to foot contour, the literature is lacking in data comparing insoles based on their material. In this randomized clinical trial, we compared the early effects of polyethylene (PE), polyurethane (PU), and carbon fiber insoles in the treatment of PF, using a set of patient-reported outcomes.

DETAILED DESCRIPTION:
Carbon fiber insoles (VKTRY, Milford, CT, USA) were initially designed to increase ground forces leading to a harder push off for faster running or higher jumping. To enable energy return, the insoles require extreme rigidity and therefore are composed of a full-length carbon-fiber base. The highly rigid construct of the carbon fiber can potentially benefit patients with plantar fasciitis by using these insoles in their own shoes, which could lead to more effective pain management, increased compliance, and improved patient outcomes. While this insole is currently being widely used by athletes, the application of this insole for PF patients has not been explored. Therefore, the aim of this study is to understand how patients respond to the these insoles compared to current standard orthotics (Superfeet Green, Superfeet Worldwide LLC. WA, USA and Aetrex L20, Aetrex Inc, NJ, USA) in a blinded randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old) with plantar fasciitis
* Adults who are competent and able to consent on their own behalf
* Patients who are seen at MGH Boston, MGH Waltham and Newton Wellesley Hospital

Exclusion Criteria:

* Patients who received an injection in the last 6 months in their plantar fascia
* Patients who will need to be treated surgically
* Patients who are non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
PROMIS-Pain interference | Baseline, 2nd-, 6th-, and 12th-week follow-ups
  measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities
PROMIS-Pain intensity | Baseline, 2nd-, 6th-, and 12th-week follow-ups
  assesses how much a person hurts. Patients are usually able to provide quantitative pain intensity estimates relatively quickly

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score | Baseline, 2nd-, 6th-, and 12th-week follow-ups
  a 42-item questionnaire with 5 subscales: pain (9 items), other symptoms (7 items), activities of daily living (ADL) (17 items), sports/recreation (5 items), and quality of life (4 items
Visual Analogue Scale for pain | Baseline, 2nd-, 6th-, and 12th-week follow-ups
  A Visual Analogue Scale (VAS) is one of the pain rating scales

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
All data acquired as specified by this protocol will be maintained and monitored by approved study staff. Approved study staff will be responsible for collecting the signed consent forms. All electronic data and subject information will be secured on non-networking password protected computers; all paperwork will be secured in locked filing cabinets. All electronic data and subject information will be secured in REDCap and will be secured on non-networking password protected computers to which only study staff will have access; all paper work will be secured in locked filing cabinets.

REFERENCES:
- [Background] Cohena-Jimenez M, Pabon-Carrasco M, Perez Belloso AJ. Comparison between customised foot orthoses and insole combined with the use of extracorporeal shock wave therapy in plantar fasciitis, medium-term follow-up results: A randomised controlled trial. Clin Rehabil. 2021 May;35(5):740-749. doi: 10.1177/0269215520976619. Epub 2020 Nov 24. PMID 33233945
- [Background] Enders, H., Vienneau, J., Tomaras, E. K., Koerger, H., Nigg, S., & Nigg, B. (2015). Soccer shoe bending stiffness significantly alters game-specific physiology in a 25-minute continuous field-based protocol. Footwear Science, 7(sup1), S91-S93. https://doi.org/10.1080/19424280.2015.1038626
- [Background] Bartolo, E., Formosa, C., & Gatt, A. (2017). The Relationship between Plantar Fasciitis and Plantar Heel Pressure. European Journal of Podiatry / Revista Europea de Podología, 3(1), 1-7. https://doi.org/10.17979/ejpod.2017.3.1.1741
- [Background] Bhimani, R., Sornsakrin, P., Vrolyk, M. A., Lubberts, B., Guss, D., DiGiovanni, C. W., & Waryasz, G. R. (2022). Use of Flexible Carbon Fiber Insoles for Hallux Rigidus: A Randomized Controlled Trial. Foot & Ankle Orthopaedics, 7(4), 2473011421S00590. https://doi.org/10.1177/2473011421S00590
- [Background] Gerrard JM, Bonanno DR, Whittaker GA, Landorf KB. Effect of different orthotic materials on plantar pressures: a systematic review. J Foot Ankle Res. 2020 Jun 11;13(1):35. doi: 10.1186/s13047-020-00401-3. PMID 32527296
- [Background] Hawke F, Burns J, Radford JA, du Toit V. Custom-made foot orthoses for the treatment of foot pain. Cochrane Database Syst Rev. 2008 Jul 16;2008(3):CD006801. doi: 10.1002/14651858.CD006801.pub2. PMID 18646168
- [Background] Lee SY, McKeon P, Hertel J. Does the use of orthoses improve self-reported pain and function measures in patients with plantar fasciitis? A meta-analysis. Phys Ther Sport. 2009 Feb;10(1):12-8. doi: 10.1016/j.ptsp.2008.09.002. Epub 2008 Nov 20. PMID 19218074